CLINICAL TRIAL: NCT02850016
Title: A Phase 2a, Randomized Study of Romidepsin With or Without 3BNC117 to Evaluate the Effects on the HIV-1 Reservoir (ROADMAP)
Brief Title: Romidepsin Plus 3BNC117 Phase 2a Study
Acronym: ROADMAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: University Hospital of Cologne (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCA-0896
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Romidepsin; 3BNC117; Broadly neutralizing antibody
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — 3BNC117 antibody; Antibodies, Monoclonal; romidepsin; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Two treatment cycles each consisting of 3BNC117 infusions (30mg/kg) + three romidepsin infusions (5mg/m2). 3BNC117 will be administered on Days 0 and 56. Romidepsin will be administered on days 2, 9, 16, 58, 65, and 72 .
  Interventions: Drug: 3BNC117; Drug: Romidepsin
- Group B (Experimental): Two treatment cycles each consisting of three romidepsin infusions (5mg/m2). Romidepsin will be administered on days 0, 7, 14, 56, 63, and 70 .
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: 3BNC117 — Intravenous Infusion of 3BNC117
  Other Names: Monoclonal Antibody
  Arms: Group A
Drug: Romidepsin — Intravenous Infusion of Romidepsin
  Other Names: HDAC inhibitor

SUMMARY:
The aim of this protocol is to evaluate the effects of romidepsin plus 3BNC117 or romidepsin alone on delaying or preventing viral rebound in ART-treated HIV-1-infected individuals during an analytical interruption of ART.

DETAILED DESCRIPTION:
This is a randomized interventional phase 2a trial of 3BNC117 and romidepsin in human immunodeficiency (HIV-1) infected patients on ART, conducted as a multi-center study at the Department of Infectious Diseases, Aarhus University Hospital, Denmark, the Rockefeller University Hospital, USA, and the University Hospital of Cologne, Germany.

Participants will be randomized 1:1 in a non-blinded fashion to receive one of two regimens:

A) Two treatment cycles each consisting of one 3BNC117 infusion (30mg/kg) + three romidepsin infusions (5mg/m2); or

B) Two treatment cycles each consisting of three romidepsin infusions (5mg/m2).

ART will be discontinued 16 weeks after the start of the second treatment cycle (analytical treatment interruption, ATI) and subjects will be monitored weekly for safety and viral rebound. The targeted enrollment is 30 subjects (15 per arm).

Leukapheresis will be performed before and after the two treatment cycles to guarantee sufficient material to investigate changes in the reservoir after the interventions.

The following criteria will require resumption of ART:

* CD4+ T cell-count <350 cells/mm³ (confirmed by repeat measurement)
* 2 consecutive plasma HIV-1 RNA measurements ≥ 200 copies/mL or above their setpoint viremia (if documented)
* Subject request
* Continued ART interruption will, in the opinion of the investigator or study advisers, pose an unacceptable risk to the subject.

If HIV-1 RNA remains undetectable at week 36, subjects will be offered to continue off ART with close monitoring, in conjunction with the subject's primary medical provider, as long as HIV-1 viral rebound does not occur. ART resumption will follow same criteria as detailed above. All subjects will be followed for a total of 48 weeks from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65 years with documented HIV-1 infection
* CD4+ T-cell count >500 cells/mm3 at screening
* On ART for a minimum of 24 months and HIV-1 RNA plasma level of < 50 copies/ml by standard assays for at least 18 months (a single viral load measurement > 50 but < 500 copies/ml during this time period is allowable).
* Individuals on protease inhibitor or NNRTI-based regimens, or regimens containing cobicistat must be willing to switch to an integrase-inhibitor-based regimen (raltegravir or dolutegravir) prior to enrollment.

Exclusion Criteria:

* Use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the investigators within the last 6 months
* Pregnancy as determined by a positive urine or serum beta-hCG.
* Participant unwilling to use two reliable contraception methods (i.e. condom with spermicide, diaphragm with spermicide, progestin-only containing intrauterine device (IUD) (eg, Mirena, Implanon, Nuva Ring), non-estrogen containing formulations of hormonal birth control drugs with condom) for the study duration.
* Currently breast-feeding.
* History of resistance to 2 or more classes of antiretroviral medications
* Any medical, psychiatric, social, or occupational condition that, as judged by the investigators, would interfere with the evaluation of study objectives (such as severe alcohol or drug abuse, dementia).
* Acute or chronic hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
* A history of AIDS-defining illness within 3 years prior to enrollment.
* History of B-cell lymphoma, including CNS lymphoma
* CD4 nadir < 200 cells/mm3
* History of significant coronary artery disease, myocardial infarction, percutaneous coronary intervention with placement of cardiac stents, or family history of sudden death at age < 50 years.
* ECG at screening that shows QTc >450 msec when calculated using the Fridericia formula from either lead V3 or V4, pathological Q-waves (Q-wave > 40 msec or depth > 0.4-0.5 mV), evidence of a ventricular pre-excitation syndromes, complete or incomplete LBBB or RBBB, second or third degree heart block, QRS duration > 120 msec, or bradycardia defined by sinus rate < 50 bps
* Use of QT-prolonging medication, renal or hepatic disease, structural heart disease or left ventricular dysfunction
* Any symptomatic or asymptomatic arrhythmia excluding sinus arrhythmia and bradycardia ≥ 50 bps.
* Laboratory abnormalities in the parameters listed below:

  1. Absolute neutrophil count ≤ 1,000 cells/μl
  2. Hemoglobin < 11 gm/dL
  3. Platelet count < 125,000 cells/μl
  4. Alanine Aminotransferase (ALT) ≥ 1.25 x ULN
  5. Aspartate Aminotransferase (AST) ≥ 1.25 x ULN
  6. Total bilirubin > 1.0 ULN
  7. Creatinine > 1.0 ULN
* Any vaccination within 14 days prior to 3BNC117 administration
* Receipt of any therapeutic HIV vaccine in the past
* Receipt of any monoclonal antibody or HDAC inhibitor of any kind in the past.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Rockefeller University
Locations (3):
- The Rockefeller University, New York, New York, United States
- Aarhus University Hospital, Aarhus, Denmark
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gruell H, Gunst JD, Cohen YZ, Pahus MH, Malin JJ, Platten M, Millard KG, Tolstrup M, Jones RB, Conce Alberto WD, Lorenzi JCC, Oliveira TY, Kummerle T, Suarez I, Unson-O'Brien C, Nogueira L, Olesen R, Ostergaard L, Nielsen H, Lehmann C, Nussenzweig MC, Fatkenheuer G, Klein F, Caskey M, Sogaard OS. Effect of 3BNC117 and romidepsin on the HIV-1 reservoir in people taking suppressive antiretroviral therapy (ROADMAP): a randomised, open-label, phase 2A trial. Lancet Microbe. 2022 Mar;3(3):e203-e214. doi: 10.1016/S2666-5247(21)00239-1. Epub 2022 Jan 24. PMID 35544074
- [Derived] Valente PK, Wu Y, Cohen YZ, Caskey M, Meyers K. Behavioral and social science research to support development of educational materials for clinical trials of broadly neutralizing antibodies for HIV treatment and prevention. Clin Trials. 2021 Feb;18(1):17-27. doi: 10.1177/1740774520948042. Epub 2020 Aug 24. PMID 32838558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 participants signed informed consent. 22 met eligibility criteria and were randomized to study groups A or B in a 1:1 ratio. 2 participants withdrew consent prior to receiving the investigational products. 20 were available for analyses.
Pre-assignment Details: Participants were screened after signing informed consent and underwent a baseline leukapheresis procedure.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 11 | 9
Completed | 10 | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants randomized to receive the interventional products
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [33 to 51] | 51 [38 to 62] | 44 [33 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 8 | 6 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
  Denmark | 3 | 2 | 5
  Germany | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Days to Viral Rebound During Analytical Treatment Interruption (ATI)
Description: Viral rebound is defined as HIV-1 RNA ≥ 200 copies/mL on 2 consecutive measurements during ATI. If viral rebound occurs, the date of the first measurement of HIV-1 RNA ≥ 200 copies/mL will be defined as "date of viral rebound
Time Frame: Week 24 to Week 36
Population: Of the 11 participants randomized to Group A, 1 chose not to interrupt ART. Of the 9 participants randomized to Group B, 1 stopped ART earlier than planned in the protocol and 1 chose not to interrupt ART.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 7
days | 18 [14 to 28] | 28 [21 to 35]

2. Secondary Outcome: Number of of Adverse Events (AE), Serious Adverse Events (SAE), and Serious Unexpected Serious Adverse Reactions (SUSAR).
Description: The occurrence of adverse events was assessed during each follow up visit. Adverse events of grades 1 or higher were reported.
Time Frame: 48 weeks
Population: All participants who received at least a single dose of the investigational products.
Measure: Number; unit: events
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 9
events
  All Adverse events related to Romidepsin | 112 | 66
  All Adverse events related to 3BNC117 | 4 | 0
  Grade 2 or higher Adverse Events Related to Romidepsin | 29 | 5
  Grade 2 or higher Adverse Events Related to 3BNC117 | 1 | 0

3. Secondary Outcome: Change in the Size of the Proviral HIV-1 Reservoir
Description: Determined by total HIV-1 DNA and episomal HIV-1 DNA (2-LTR) in circulating total CD4+ T cells at baseline and prior to the ATI period (week 24).
Time Frame: baseline and week 24
Population: Participants who completed dosing per protocol and underwent leukapheresis at baseline and following the interventions (week 24).
Measure: Median (Inter-Quartile Range); unit: HIV-1 DNA per million CD4+ T cells
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 9
HIV-1 DNA per million CD4+ T cells | 58 [27 to 482] | 46 [0 to 270]

4. Secondary Outcome: Plasma HIV-1 RNA
Description: As measured by a routine clinical assay (Cobas Taqman; detection limit 20 copies/mL), a transcription mediated amplification (TMA)-based assay (detection limit 12 copies/ml) and/or a single copy assay (detection limit 1-2 copies/mL)
Time Frame: 48 weeks
Population: Participants with detectable plasma HIV-1RNA during the treatment cycles measure by commercial assays.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 9
Participants | 4 | 4

5. Other Pre Specified Outcome: HIV-1 Transcriptional Activity as Determined by Unspliced HIV-1 RNA (CA usHIV-1 RNA) in Circulating Total CD4+ T Cells.
Description: The median fold-change in cell-associated unspliced HIV-1 RNA concentrations after romidepsin administration across all infusions
Time Frame: baseline and week 24
Population: Participants who completed dosing according to protocol.
Measure: Median (Inter-Quartile Range); unit: CA-us HIV-1 RNA per million CD4 T cells
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 9
CA-us HIV-1 RNA per million CD4 T cells | 9 [1 to 111] | 11 [5 to 85]

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: The definition of adverse event and/or serious adverse event DO NOT differ from the clinicaltrials.gov definitions
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 11/11 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=11) | Group B (N=9)
Nausea (Gastrointestinal disorders) | 11 (29) | 9 (9)
Headache (General disorders) | 4 (13) | 3 (10)
Fatigue (General disorders) | 5 (12) | 4 (4)
Chills (General disorders) | 3 (8) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (8) | 2 (2)
Decreased phosphorus (Investigations) | 1 (5) | 2 (5)
Malaise (General disorders) | 3 (5) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (3) | 0 (0)
Increased creatinine (Renal and urinary disorders) | 2 (3) | 0 (0)
Xerostomia (Eye disorders) | 3 (3) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3)
Neutropenia (Cardiac disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Prolonged QT interval (Cardiac disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02850016/Prot_SAP_000.pdf